CLINICAL TRIAL: NCT03696225
Title: Assessment and Treatment of Cognitive Functioning Deficits in Veterans With PTSD
Acronym: CCTPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2762-W; 1IK2RX002762-01A1 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Cognitive Function
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a parallel randomized controlled pilot trial.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be masked to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compensatory Cognitive Training (CCT) (Experimental): Compensatory Cognitive Training draws from the theoretical literature on compensatory strategy training for other cognitively impaired populations (e.g., Huckans et al., 2013; Twamley et al., 2010; Storzbach et al., 2016). It is a rehabilitation model that aims to teach individuals strategies that allow them to work around cognitive deficits. Consistent with this model and the expert recommendations for civilians and Service members with TBI (Cicerone, 2011), manualized CCT treatment provides training in compensatory attention and learning/memory skills, formal problem-solving strategies applied to daily problems, and the use of external aids such as calendar systems and assistive devices to promote completion of daily tasks (Storzbach et al., 2016).
  Interventions: Behavioral: Compensatory Cognitive Training (CCT)
- Treatment as Usual (TAU) (Active Comparator): All TAU participants have an ongoing VA mental health provider and received ongoing mental health care during the course of the study (generally weekly individual or group sessions focusing on evidence-based PTSD treatment).
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Compensatory Cognitive Training (CCT) — Compensatory Cognitive Training draws from the theoretical literature on compensatory strategy training for other cognitively impaired populations (e.g., Huckans et al., 2013; Twamley et al., 2010; Storzbach et al., 2016). It is a rehabilitation model that aims to teach individuals strategies that allow them to work around cognitive deficits. Consistent with this model and the expert recommendations for civilians and Service members with TBI (Cicerone, 2011), manualized CCT treatment provides training in compensatory attention and learning/memory skills, formal problem-solving strategies applied to daily problems, and the use of external aids such as calendar systems and assistive devices to promote completion of daily tasks (Storzbach et al., 2016).
  Other Names: CCT
  Arms: Compensatory Cognitive Training (CCT)
Behavioral: Treatment as Usual (TAU) — All TAU participants have an ongoing VA mental health provider and received ongoing mental health care during the course of the study (generally weekly individual or group sessions focusing on evidence-based PTSD treatment).
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
Approximately half a million Veterans receiving services at the VA have Posttraumatic Stress Disorder (PTSD). PTSD is strongly associated with cognitive functioning deficits in areas of concentration, attention, memory, learning, verbal abilities, processing speed, and multitasking. Compensatory Cognitive Training (CCT) is an evidence-based intervention for cognitive problems that is effective in other Veteran populations such as those with a history of traumatic brain injury (TBI), but CCT has not yet been tested in Veterans with PTSD who don't have a history of TBI. The investigators will conduct a pilot randomized controlled trial (RCT) of CCT in Veterans who have been treated for PTSD but continue to have cognitive functioning deficits. The investigators will examine feasibility, acceptability, participant characteristics, and effect size estimates in preparation for a fully-powered RCT of CCT for PTSD-related cognitive functioning deficits.

DETAILED DESCRIPTION:
Project Background: PTSD is associated with deficits in cognitive functioning including memory, learning, processing speed, concentration, attention, and executive functioning. Though many Veterans benefit from evidence-based psychotherapy (EBP) for PTSD, many Veterans have cognitive functioning deficits even after completing EBP for PTSD. There are no evidence-based treatments for these Veterans. Compensatory Cognitive Training (CCT) is improves cognitive functioning in Veterans with brain injury history, but is not yet tested in Veterans with PTSD.

Project Aims: This study will evaluate feasibility, acceptability, and participant characteristics, and estimate effect sizes, in a pilot test of CCT for Veterans with PTSD-related cognitive problems. Data from this study will form the basis for a future, fully powered trial testing the effectiveness of CCT for cognitive problems in Veterans with PTSD.

Project Methods: The investigators will recruit Veterans from local VA mental health clinics, using the VA's Corporate Data Warehouse (CDW) to identify potentially eligible Veterans if needed. The investigators will compare CCT vs. treatment as usual for 36 Veterans with PTSD-related cognitive functioning deficits. The investigators will calculate rates of recruitment, retention, and intervention participation. Statistical significance will be examined, though the investigators' focus will be on effect size estimates, score ranges, and variability to plan for a follow-up, fully powered RCT.

Anticipated Impact: PTSD-related cognitive functioning deficits are a significant problem for many Veterans. CCT is an effective cognitive rehabilitation intervention for Veterans with a history of brain injury, but VA clinicians need data on its effectiveness for Veterans with PTSD-related cognitive functioning deficits. These studies will provide the data necessary for a larger scale RCT proposal if results show that CCT is as promising as expected for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Veterans must meet Diagnostic and Statistical Manual 5 (DSM-5) criteria for PTSD with evidence-based PTSD treatment participation within the past 2 years.
* Must have an individual mental health provider/case manager assigned for coordination of care and management of crises as well as provision of treatment as usual if Veteran is randomly assigned to this condition.
* Report subjective cognitive complaints, such as problems with memory, attention/concentration, and executive function (e.g., planning, organization, problem-solving, decision-making).
* Referring provider observes mild cognitive problems that interfere with daily life (e.g., forgetting appointments or medications, poor performance at work or school, difficulty remembering information, trouble focusing in treatment sessions, trouble following through on goals).
* Fluent English speaker.
* Able to read and write and provide informed consent.

Exclusion Criteria:

* No history of traumatic brain injury (tbi) of any severity or another major medical condition likely to significantly impact cognitive functioning such as stroke, multiple sclerosis (MS), Parkinson's, or a brain tumor.
* Do not meet criteria for bipolar disorder or a psychotic disorder. Do not have a diagnosis of a substance dependence disorder within the past 30 days.
* Do not have active suicidal intent indicating significant clinical risk (which would suggest that a treatment targeting suicidal intent is indicated).
* Cognitive problems are not severe (i.e., no dementia). Cognitive problems do NOT interfere with a Veteran's overall ability to live independently or care for him/herself.
* Not currently participating in any type of brain stimulation treatment.
* No significant auditory/visual impairments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Elin O'Neil, PhD MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Started | 13 | 8
Completed | 10 | 6
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12.89) | 45.63 (14.3) | 45.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 13 | 4 | 17
  Non-Hispanic Black | 0 | 2 | 2
  Native American | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 8 | 21
Education (years) [Mean (Standard Deviation); unit: years] | 14.31 (1.93) | 15.75 (2.44) | 14.86 (2.20)
Mental Health Diagnosis [Count of Participants; unit: Participants]
  PTSD | 13 | 6 | 19
  Major Depressive Disorder | 7 | 4 | 11
  Panic Disorder | 5 | 1 | 6
  Agoraphobia | 9 | 3 | 12
  Social Anxiety | 5 | 2 | 7
  Generalized Anxiety Disorder | 5 | 1 | 6
  Alcohol Use Disorder | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Prospective-Retrospective Memory Questionnaire (PRMQ; Crawford et al., 2006)
Description: Self-report severity measure of prospective (remembering to do something in the future) and retrospective (remembering something from the past) memory problems relevant to every day life. Higher scores represent worse outcomes. Total score ranges from 0-64.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a scale
  Baseline | 50.38 (10.145) | 38.5 (15.875)
  3-Month: number analyzed (Participants) | 8 | 4
  3-Month | 47.875 (9.96) | 42.5 (16.01)
  6-Month: number analyzed (Participants) | 5 | 7
  6-Month | 39.8 (13.846) | 45.857 (16.406)

2. Primary Outcome: Multiple Sclerosis Neuropsychological Screening Questionnaire - Patient Version (MSNQ; Benedict et al., 2003)
Description: Self-report severity measure of attention and organizational problems. Scores on the MSNQ range from 0 to 58, with higher scores indicating greater cognitive impairment.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a scale
  Baseline | 33.15 (8.143) | 22.75 (12.903)
  3-Month: number analyzed (Participants) | 8 | 4
  3-Month | 29.375 (7.52) | 26.5 (11.387)
  6-Month: number analyzed (Participants) | 5 | 6
  6-Month | 22.6 (14.117) | 29.833 (14.442)

3. Primary Outcome: California Verbal Learning Test (CVLT-II; Delis et al., 2000)
Description: Comprehensive measurement of verbal learning and memory and includes a forced choice validity. The total raw score is the sum of correct responses on the five presentations; scores range from 0-80. Higher scores represent better outcomes.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a measure
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a measure
  Baseline | 52.77 (11.047) | 52.88 (10.602)
  3-Month: number analyzed (Participants) | 10 | 6
  3-Month | 62.8 (8.066) | 58.33 (16.207)
  6-Month: number analyzed (Participants) | 3 | 7
  6-Month | 52.333 (9.713) | 63.857 (14.622)

4. Primary Outcome: Wechsler Adult Intelligence Scale (WAIS-IV) Coding Subtest (Wechsler, 2008)
Description: A measure of processing speed. Higher scores represent better outcomes. Scores range from 0-155.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a measure
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a measure
  Baseline | 69.38 (12.646) | 73.25 (9.910)
  3-Month: number analyzed (Participants) | 8 | 4
  3-Month | 77 (17.171) | 79.25 (16.008)
  6-Months: number analyzed (Participants) | 1 | 7
  6-Months | 88.00 (0.00) | 75.143 (13.184)

5. Primary Outcome: Controlled Oral Word Association Test (Benton, Hamsher, & Sivan, 1983)
Description: The Controlled Oral Word Association (COWA) Test measures word generation, verbal fluency, and executive functioning. Participants are asked to name as many words as they can starting with a specific letter (i.e., F, A, S) within one minute, and as many words as possible in a specified category (i.e., animals) within one minute. Total score is the sum of responses (three letter trials, one category trial). Higher scores represent better outcomes. Total score ranges are affected by age and education.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
Number of words
  Letters - Baseline | 42.69 (11.828) | 44.75 (11.829)
  Categories - Baseline | 24.38 (6.423) | 27.0 (5.210)
  Letters - 3-Months: number analyzed (Participants) | 9 | 7
  Letters - 3-Months | 40.00 (14.169) | 46.0 (10.017)
  Categories - 3-Months: number analyzed (Participants) | 9 | 7
  Categories - 3-Months | 22.667 (6.614) | 21.143 (6.669)
  Letters - 6-Months: number analyzed (Participants) | 3 | 7
  Letters - 6-Months | 47.000 (12.288) | 48.571 (11.559)
  Categories - 6-Months: number analyzed (Participants) | 3 | 7
  Categories - 6-Months | 23.667 (3.786) | 23.429 (3.101)

6. Primary Outcome: Halstead Reitan Trailmaking Test (Trails A & B; Reitan & Wolfson, 1985)
Description: Measures visual tracking, processing speed, and executive functioning. Scores represent the amount of time to complete the task (in seconds), range from 10-366, and higher numbers represent worse outcomes.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
Seconds
  Trails A - Baseline | 26.62 (4.840) | 22.50 (9.071)
  Trails B - Baseline | 58.85 (12.089) | 50.63 (10.542)
  Trails A - 3-Month: number analyzed (Participants) | 8 | 4
  Trails A - 3-Month | 22.125 (6.999) | 20.0 (6.481)
  Trails B - 3-Month: number analyzed (Participants) | 8 | 4
  Trails B - 3-Month | 46.5 (9.15) | 45.0 (15.663)
  Trails A - 6-Month: number analyzed (Participants) | 1 | 7
  Trails A - 6-Month | 12.0 (0) | 20.571 (6.554)
  Trails B - 6-Month: number analyzed (Participants) | 1 | 7
  Trails B - 6-Month | 38.0 (0) | 45.286 (9.411)

7. Primary Outcome: World Health Organization Disability Assessment Scale (WHODAS 2.0)
Description: Self-report measure of quality of life and global functioning. Higher scores represent worse outcomes. Total score ranges from 0-144.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 11 | 8
score on a scale
  Baseline | 63.727 (22.136) | 43.125 (26.167)
  3-Month: number analyzed (Participants) | 7 | 4
  3-Month | 51.286 (27.066) | 42.5 (40.435)
  6-Month: number analyzed (Participants) | 5 | 5
  6-Month | 65.4 (43.964) | 52.6 (15.534)

8. Primary Outcome: Quality of Life in Neurological Disorders (Neuro-QOL): Cognitive, Ability to Participate in Social Roles and Activities, and Sleep Scales
Description: Self-report measure of quality of life, cognitive functioning, sleep functioning, and social functioning. Higher scores represent lower functioning. Total scores range from 52 to 260.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
scores on a scale
  Baseline | 76.00 (16.703) | 99.88 (31.904)
  3-Months: number analyzed (Participants) | 8 | 4
  3-Months | 88.375 (19.175) | 92.00 (43.772)
  6-Months: number analyzed (Participants) | 5 | 7
  6-Months | 100.6 (30.867) | 92.857 (27.267)

9. Primary Outcome: Memory Compensation Questionnaire (MCQ; de Frias & Dixon, 2005)
Description: A 44-item self-report questionnaire that rates the extent of use of various strategies to improve memory performance relevant to daily living. Higher scores represent better outcomes. Total score ranges from 0-176.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a scale
  Baseline | 105.38 (26.943) | 101.88 (30.954)
  3-Month: number analyzed (Participants) | 8 | 4
  3-Month | 91.125 (22.106) | 86.25 (47.528)
  6-Month: number analyzed (Participants) | 5 | 7
  6-Month | 104.4 (48.190) | 91.143 (38.507)

10. Primary Outcome: Portland Cognitive Strategies Scale 2.0 (PCSS)
Description: Measures compensatory cognitive strategy use through two scales; how often skills are used and how useful. Higher scores represent more skill use and more perceived usefulness. Total score ranges from 0-60 per scale.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a scale
  Often - Baseline | 36.46 (14.033) | 45.88 (8.202)
  Useful - Baseline | 29.42 (5.915) | 33.63 (4.984)
  Often - 3-Months: number analyzed (Participants) | 11 | 6
  Often - 3-Months | 31.182 (21.042) | 31.167 (21.170)
  Useful - 3-Months: number analyzed (Participants) | 8 | 4
  Useful - 3-Months | 30.875 (2.800) | 29.00 (2.708)
  Often - 6-Months: number analyzed (Participants) | 5 | 6
  Often - 6-Months | 45.0 (9.823) | 44.833 (8.565)
  Useful - 6-Months: number analyzed (Participants) | 5 | 6
  Useful - 6-Months | 32.8 (4.087) | 30.833 (4.446)

11. Primary Outcome: Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span Subtest (Wechsler, 2008)
Description: Measures attention, working memory, processing speed, and reliable digit span validity. Higher scores represent better outcomes. Scores on each subtest (forward, backward, and sequential) range from 0-16 and are reported as WAIS Scaled Scores. Total score (range 0-48) is the sum of each subtest.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a measure
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a measure
  Baseline | 27.62 (3.664) | 28.88 (6.728)
  3-Months: number analyzed (Participants) | 10 | 6
  3-Months | 29.4 (4.858) | 32.33 (1.21)
  6-Months: number analyzed (Participants) | 3 | 7
  6-Months | 32.0 (6.557) | 31.571 (4.577)

12. Secondary Outcome: PTSD Checklist (PCL-5; Weathers et al., 2013)
Description: PTSD symptoms and severity. Higher scores indicates more severe symptomology. Total score ranges from 0-80.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
score on a scale
  Baseline | 41.31 (18.287) | 34.75 (24.259)
  3-Months: number analyzed (Participants) | 8 | 3
  3-Months | 36.375 (16.792) | 20.0 (27.785)
  6-Months: number analyzed (Participants) | 5 | 7
  6-Months | 29.0 (23.548) | 34.571 (19.890)

13. Secondary Outcome: Patient Health Questionnaire (PHQ-9; Spitzer, Kroenke, & Williams, 1999)
Description: A brief, nine-item depression assessment questionnaire used to screen for depression and monitor its severity. Higher scores represent worse outcomes. Total score ranges from 0-27.
Time Frame: change from baseline to 3 and 6 months
Population: Due to drop-out and COVID precautions, there were less participants who completed measures at 3- and 6-Month follow-ups
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 8
Score on a scale
  Baseline | 22.23 (8.228) | 22.25 (9.573)
  3-Months: number analyzed (Participants) | 8 | 4
  3-Months | 19.5 (5.155) | 19.0 (10.424)
  6-Months: number analyzed (Participants) | 5 | 7
  6-Months | 19.4 (7.127) | 21.571 (7.743)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Compensatory Cognitive Training (CCT) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Coronavirus disease shutdown resulted in less recruitment than initially anticipated. Groups and assessments were moved to a remote, phone-based format which may have limited understanding and application of skills taught in groups. Exclusion criteria included some diagnoses (i.e., history of TBI) which are frequently comorbid with PTSD, which limited the sample and affected recruitment efforts. Low demographic variability limits representation and generalizability to the larger population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03696225/Prot_SAP_000.pdf